CLINICAL TRIAL: NCT07357597
Title: A Phase IV, Open-Label, Single-Arm Study of Prophylaxis for Datopotamab Deruxtecan-related Stomatitis in Eligible Patients With Metastatic or Inoperable Locally Recurrent Breast Cancer or Locally Advanced or Metastatic Epidermal Growth Factor Receptor-Mutated Non-Small Cell Lung Cancer (TROPION-SWISH)
Brief Title: An Open-label, Single-arm Study of Prophylaxis for Datopotamab Deruxtecan (Dato-DXd) -Related Stomatitis in Eligible Patients With Metastatic or Inoperable Locally Recurrent Breast Cancer or Locally Advanced or Metastatic Epidermal Growth Factor Receptor-Mutated Non-small Cell Lung Cancer.
Acronym: TROPION-SWISH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D926UL00001
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Stomatitis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexamethasone 0.5 mg/5 mL Mouthwash (Experimental): Participants will use dexamethasone 0.5 mg/5 mL alcohol-free mouthwash (10 mL, 4 times daily, swish for approximately 2 minutes, then spit out without swallowing).
  Participants will remain without food or drink for at least 30 minutes after use of dexamethasone
  Interventions: Drug: Dexamethasone mouthwash; Drug: Datopotamab Deruxtecan (Dato-DXd)

INTERVENTIONS:
Drug: Dexamethasone mouthwash — Dexamethasone steroid-based oral solution, comprised of 0.5 milligrams per 5mL of alcohol-free dexamethasone.
Drug: Datopotamab Deruxtecan (Dato-DXd) — Commercially available Dato-DXd is prescribed and administered to participants according to standard of care
  Other Names: Datroway

SUMMARY:
This is a multicenter, open-label, single-arm study of prophylaxis for Dato-DXd-related stomatitis in eligible patients with metastatic or inoperable locally recurrent breast cancer or locally advanced or metastatic Epidermal Growth Factor Receptor-Mutated (EGFRm) non-small cell lung cancer.

DETAILED DESCRIPTION:
The purpose of this Phase IV study is to describe the incidence and severity of Dato-DXd treatment-emergent grade ≥ 2 stomatitis in participants receiving prophylactic dexamethasone mouthwash within the first 12 weeks of study treatment (ie, Dato-DXd dosing).

The study will enroll an estimated 100 participants across approximately 35 sites in the U.S. Enrollment of participants is planned to occur over approximately 18 months, with a minimum of 12 weeks of follow-up for each participant after the first Dato-DXd dose.

This study has one arm, and the study population will consist of 2 independent cohorts (approximately 50 participants in each cohort):

* Breast cohort (Cohort 1)
* Lung cohort (Cohort 2)

Participants will receive the study intervention, dexamethasone mouthwash, throughout the duration of their standard of care treatment with Dato-DXd.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all the following criteria apply:

Disease Characteristics

1. Patients with any of the following disease characteristics are eligible (specific population subject to FDA Dato-DXd label):

   • Patients with unresectable or metastatic HR+/HER2- (IHC 0, IHC 1+, or IHC 2+/ISH-) breast cancer who have received prior ET and chemotherapy for unresectable or metastatic disease.

   OR

   • Adult patients with unresectable or metastatic TNBC who are not candidates for PD-1/PD-L1 inhibitor therapy. Participants will be enrolled upon FDA approval on use of Dato-DXd for this indication.

   OR

   • Patients with locally advanced or metastatic EGFRm NSCLC who have received prior EGFR-directed therapy and platinum-based chemotherapy.

   Age
2. Patient must be ≥ 18 years, at the time of signing the informed consent.

   Type of Patient and Disease Characteristics-
3. Has documentation that Dato-DXd will be prescribed for the labelled indication and has not received any dose of Dato-DXd prior to enrollment.
4. Is willing to comply with use of prophylactic dexamethasone mouthwash at the start of first infusion and throughout Dato-DXd administration.
5. ECOG performance status 0 or 1.
6. Has adequate bone marrow function (hemoglobin ≥ 9 g/dL; red blood cell/plasma transfusion is not allowed within 1 week prior to screening assessment).
7. All women of childbearing potential must have a negative serum pregnancy test result at screening.

   Informed Consent
8. Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the ICF and the protocol.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply:

1. Has received Dato-DXd prior to enrollment.

   Medical Conditions
2. As judged by the investigator, any evidence of cardiac, pulmonary, vascular, and other renal conditions which in the investigator's opinion makes it undesirable for the patient to participate in the study.
3. Has any-grade active and uncontrolled stomatitis or mouth ulcers at baseline (participants with prior medical history of stomatitis or mouth ulcers are eligible).
4. Use of steroid-containing mouthwash is contraindicated in, including but not limited to:

   * Active oral infections (eg, viral, bacterial, or fungal), where the use of a steroid-containing mouthwash may impair local immune response and delay healing
   * Known hypersensitivity or allergy to corticosteroids or any excipients contained in the mouthwash formulation
5. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals; suspected infections (eg, prodromal symptoms); or inability to rule out infections (participants with localized fungal infections of skin or nails are eligible).
6. Has clinically significant corneal disease.
7. Has a history of severe hypersensitivity reactions to either the drug or inactive ingredients of Dato-DXd (including, but not limited to, polysorbate 80).
8. Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
9. Is pregnant, or breastfeeding, or planning to become pregnant.

   Other Exclusions
10. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
11. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
12. Previous enrollment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Dato-DXd treatment-emergent grade ≥ 2 stomatitis in patients receiving prophylactic dexamethasone mouthwash within first 12 weeks of study treatment | From date of first dose of study treatment until 12 weeks after date of first dose of study treatment
  Incidence is defined as the proportion of participants who develop National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 grade ≥ 2 stomatitis accompanied by either a Normalcy of Diet Subscale score ≤ 50 and/or a Numeric Rating Scale (NRS) oral-pain score of 7 on 2 consecutive days or 8, 9, or 10 on any one day.
  Severity will be based on the highest NCI-CTCAE v5.0 grade of stomatitis experienced by each participant.
  CTCAE displays Grades 1-5 with descriptions of severity for each adverse event (AE). Grade 1 for mild symptoms and Grade 5 for death related to AE.
  The Normalcy of Diet Subscale assesses the degree to which a patient can eat a normal diet and drink liquids. The scale is a ranking of 10 food categories, from easy-to-eat to difficult-to-eat.
  The Numeric Rating Scale is a scale for self-reporting of pain. Scores range from 0-10, with higher scores meaning the worst pain possible (0=no pain to 10=worst possible pain).

SECONDARY OUTCOMES:
Incidence and severity of Dato-DXd treatment-emergent grade ≥ 2 stomatitis | From date of first dose of study treatment until 6 and 9 weeks after date of first dose of study treatment
  This will be determined using the composite stomatitis definition in the primary outcome. Will be repeated within 6 weeks and within 9 weeks of study treatment.
Incidence and severity of treatment-emergent stomatitis overall, by maximum CTCAE grade, and CTCAE grade ≥ 2 | From date of first dose of study treatment until 6, 9 and 12 weeks after date of first dose of study treatment
  This will be determined using stomatitis CTCAE grade only. Will be analysed at 6, 9 and 12 weeks.
Time to onset of grade ≥ 2 stomatitis | From date of first dose until earliest of diagnosis of grade ≥2 stomatitis, Dato-DXD discontinuation and death, whichever occurs first, assessed up to approximately 21 months
  The time (in days) from the date of the first dose of Dato-DXd to the date of first onset to a grade ≥ 2 stomatitis event. The measure of primary interest is median time to onset.
Time to resolution of Dato-DXd-related grade ≥ 2 stomatitis | From date of diagnosis of grade ≥2 stomatitis until the earliest date of event resolved or reduced in severity to grade 1, assessed up to approximately 21 months
  Number of days from the date of onset of stomatitis grade ≥ 2 until the earliest date of event resolved or reduced in severity to grade 1. The measure of primary interest is median time to resolution.
Proportion of participants with a dose modification for Dato-DXd due to stomatitis | From date of first dose until earliest of Dato-DXD discontinuation and death, assessed up to approximately 21 months
  Dose modification is defined as dose reduction, delay, or discontinuation due to stomatitis Treatment-Emergent Adverse Event (TEAE).
Participant adherence to dexamethasone mouthwash | From date of first dose of study treatment until 12 weeks after date of first dose of study treatment
  Adherence to dexamethasone mouthwash will be assessed by cohort using the Daily Activities Diary. The measure of primary interest is the median number of swished mouthwashes per day.
Safety and tolerability of Dato-DXd in participants receiving prophylactic dexamethasone mouthwash | From date of first dose of study intervention until 28 days after the last dose (Safety Follow-up), approximately 21 months
  Safety and tolerability will be evaluated by cohort in terms of AEs (graded by NCI-CTCAE v5.0) and in terms of the following:
  * Incidence and severity of TEAEs and Serious Adverse Events (SAEs), including oral infections (such as fungal infections) associated with the use of the dexamethasone mouthwash
  * Eastern Cooperative Oncology Group (ECOG) performance status
  * Vital signs and physical examination
  * Clinical chemistry, hematology, urinalysis, and coagulation assessments
  * Use of antifungal medication for treating dexamethasone-related fungal infection.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Duarte, California
  - Research Site, Glendale, California
  - Research Site, Lakewood, California
  - Research Site, Torrance, California
  - Research Site, Athens, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, Reno, Nevada
  - Research Site, Westbury, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, Fairfax, Virginia
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org